CLINICAL TRIAL: NCT05859789
Title: EFFECT OF MEDITERRANEAN DIET ON SEXUAL FUNCTION IN WOMEN WITH METABOLIC SYNDROME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sara Magdy Ahmed, PRINCIPAL INVESTIGATOR, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004338
Record Dates: First submitted 2023-05-05; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Metabolic Syndrome in Women

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group: Kegel exercise group (Active Comparator): will receive Kegel exercise (3 sessions /week for 12 weeks)- Each female will be asked to "Try to squeeze her pelvic floor muscles as much as possible". She was instructed that the numbers she saw at the top of screen indicated the activity of the muscle (electrical activity), in microvolt (mv).
  * The therapeutic session will be repeated 3 sessions /week for 12 weeks for each female in both groups (A&B).
  * Each female will be instructed to Tighten her pelvic floor muscles. Hold tight and count 3 to 5 seconds, relax the muscles and count 3 to 5 seconds, then repeat 10 times, 3 times a day at least three sets of 10 to 15 repetitions a day as a home program
  * They will be instructed not to use abdomen, thighs or buttock muscles during the contraction, avoid holding breath. Instead, breathe freely during the exercises.
  Interventions: Procedure: kegel exercise
- study group: Kegel exercise combined with Mediterranean diet regimen for 12 weeks. (Experimental): kegel and Mediterranean diet regimen :kegel ex same as controlled group in addition toMediterranean diet. The recommended composition of the dietary regimen was the following: carbohydrates 50-60%, proteins 15-20%, total fat o30%, saturated fat 10% and less than 300 mg of cholesterol consumed per day. Moreover, subjects Will
  Interventions: Procedure: kegel exercise; Other: Mediterranean diet regimen for 12 weeks.

INTERVENTIONS:
Procedure: kegel exercise — * Each female will be asked to "Try to squeeze her pelvic floor muscles as much as possible". She was instructed that the numbers she saw at the top of screen indicated the activity of the muscle (electrical activity), in microvolt (mv).
  * The therapeutic session will be repeated 3 sessions /week for 12 weeks for each female in both groups (A&B).
  * Each female will be instructed to Tighten her pelvic floor muscles. Hold tight and count 3 to 5 seconds, relax the muscles and count 3 to 5 seconds, then repeat 10 times, 3 times a day at least three sets of 10 to 15 repetitions a day as a home program
  * They will be instructed not to use abdomen, thighs or buttock muscles during the contraction, avoid holding breath. Instead, breathe freely during the exercises.
Other: Mediterranean diet regimen for 12 weeks. — kegel ex in addition to mediterrian diet . The recommended composition of the dietary regimen was the following: carbohydrates 50-60%, proteins 15-20%, total fat o30%, saturated fat 10% and less than 300 mg of cholesterol consumed per day. Moreover, subjects Will be advised to consume at least 250-300 g of fruits, 125-150 g of vegetables and 25-50 g of nuts per day.
  Arms: study group: Kegel exercise combined with Mediterranean diet regimen for 12 weeks.

SUMMARY:
Metabolic syndrome (MS) is a cluster of metabolic abnormalities that includes hypertension, central obesity, insulin resistance, type 2-diabetes and atherogenic dyslipidaemia (1). A woman's sexual health is associated with several psychological and interpersonal factors, and may be affected by aging and metabolic changes (2).

Obesity, hypertension, dyslipidemia, and type 2-diabetes which are conditions frequently present in women with metabolic syndrome are considered risk factors for atherosclerosis and endothelial dysfunction which impairs tissue oxygenation and causes subsequent functional and structural damage to the female genital tract. A decrease in pelvic blood flow secondary to atherosclerotic disease leads to fibrosis of the vaginal wall and clitoral smooth muscle, eventually resulting in vaginal dryness and dyspareunia (3).

Women with metabolic syndrome showed higher prevalence of sexual inactivity and low sexual desire, orgasm, satisfaction, and Female sexual function (FSFI) total score in respect to women without metabolic syndrome (4). There is a link between diet and sexual performance markers to get and maintain lubrication, orgasm, and frequency of sex, as food has a favourable or negative impact on sexual activity for both sexes at any age (5). The Mediterranean diet (Med Diet) is one of the most widely described and evaluated dietary patterns in scientific literature. It is based on the traditional foods that people used to eat in countries bordering the Mediterranean Sea, including France, Spain, Greece, and Italy. It is characterized by high intakes of vegetables, legumes, fruits, nuts, grains, fish, seafood, extra virgin olive oil, and a moderate intake of red wine (6). Previous studies proved that Kegel exercise raise the level of sexual satisfaction, as the pelvic floor muscle (PFM) specifically the pubococcygeus and iliococcygeus muscles are responsible for the rhythmic involuntary contractions during orgasm (7).

According to the authors' knowledge, no prior research studied the effect of Mediterranean diet on sexual function in women with metabolic syndrome.

DETAILED DESCRIPTION:
200 patients with metabolic syndrome complaining of sexual dysfunction, aged 25-40 years, were randomized into two equal groups, the control group (A) received sessions of Kegel exercise three times per week for 12 weeks, the study group (B) received Kegel exercise combined with Mediterranean diet regimen for 12 weeks. Female sexual function index (FSFI) questionnaire was used to evaluate sexual function of each woman in both groups, while sexual quality of life-female (SQOL_F) questionnaire was used to assess quality of life (QoL) of each woman in both groups before and after treatment.

All women will be included in this study if they fulfill the following criteria:

1. Sexually active women diagnosed with metabolic syndrome and complaining of sexual dysfunction:

   * Abdominal adiposity (waist circumference is >88 cm)
   * Low serum high density lipoprotein cholesterol
   * Hypertriglyceridemia (elevated triglyceride of >150 mg/dl)
   * Elevated blood pressure >130/85mmHg
   * Abnormal glucose homeostasis (fasting plasma glucose concentration is >110mg/dl).
2. Their age will range (25- 35 ) years
3. Body mass index (BMI) ≥ (25-30) kg/m2.

Women who had met one of the following criteria will be excluded from the study:

* Women has cardiovascular disease
* Psychiatric problems
* History of alcohol abuse
* Smoker women
* Taking medication

ELIGIBILITY:
Inclusion Criteria:All women will be included in this study if they fulfill the following criteria:

1. Sexually active women diagnosed with metabolic syndrome and complaining of sexual dysfunction:

   * Abdominal adiposity (waist circumference is >88 cm)
   * Low serum high density lipoprotein cholesterol
   * Hypertriglyceridemia (elevated triglyceride of >150 mg/dl)
   * Elevated blood pressure >130/85mmHg
   * Abnormal glucose homeostasis (fasting plasma glucose concentration is >110mg/dl).
2. Their age will range (25- 35 ) years
3. Body mass index (BMI) ≥ (25-30) kg/m2.

   -

   Exclusion Criteria:

   Women who had met one of the following criteria will be excluded from the study:
   * Women has cardiovascular disease
   * Psychiatric problems
   * History of alcohol abuse
   * Smoker women
   * Taking medication

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 200 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Female sexual function index (FSFI) questionnaire | up to 12 weeks
Sexual Quality of Life Questionnaire- Female | up to 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Egypt , Giza, Giza, Egypt